CLINICAL TRIAL: NCT00689117
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Active And Vehicle-Controlled Study Of The Safety And Efficacy Of CT Gel in Subjects With Acne Vulgaris
Brief Title: A Clinical Study to Evaluate the Safety and Effectiveness of an Investigational Product Called CT Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114681; W0265-03 (Other: Stiefel)
Record Dates: First submitted 2008-05-24; First posted 2008-06-03 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris; Acne
Keywords: Acne Vulgaris; Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Tretinoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): CT Gel
  Interventions: Drug: CT Gel
- 2 (Active Comparator): Clindamycin Gel (clindamycin)
  Interventions: Drug: Clindamycin Gel (clindamycin )
- 3 (Active Comparator): Tretinoin Gel (tretinoin)
  Interventions: Drug: Tretinoin Gel (tretinoin)
- 4 (Placebo Comparator): Vehicle Gel
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: CT Gel — Topical gel consisting of clindamycin 1% and tretinoin 0.025%, applied once daily in the evening for 12 weeks
  Arms: 1
Drug: Clindamycin Gel (clindamycin ) — Clindamycin 1% gel applied topically once daily in the evening for 12 weeks
  Arms: 2
Drug: Tretinoin Gel (tretinoin) — Tretinoin 0.025% gel applied topically once daily in the evening for 12 weeks
  Arms: 3
Drug: Vehicle Gel — Topical gel without clindamycin or tretinoin applied topically once daily in the evening for 12 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of CT Gel in subjects with acne vulgaris. The hypothesis is that CT Gel is superior to Clindamycin Gel, Tretinoin Gel and Vehicle Gel for the treatment of acne vulgaris.

DETAILED DESCRIPTION:
CT Gel is a fixed-combination product that addresses the multifactorial factors of acne vulgaris pathogenesis. Based on numerous nonclinical pharmacology studies of each active ingredient, it is expected that this new product will have three biological actions: 1) comedolytic, 2) antimicrobial, and 3) anti-inflammatory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 12 years of age or older in good general health
* Investigator's Static Global Assessment (ISGA) score of 2 or greater at Baseline

Exclusion Criteria:

* Any nodulo-cystic lesions at Baseline
* Pregnancy or breast feeding
* History or presence of regional enteritis or inflammatory bowel disease or similar symptoms.
* Treatment with estrogens, including oral, implanted and topical contraceptives, androgens, or anti-androgenic agents for 12 weeks or less prior to study start.
* Use of topical anti-acne medications within the past 2 weeks.
* Use of topical or systemic antibiotics on the face within the past 2 weeks.
* Use of topical or systemic corticosteroids within the past 2 weeks.
* Use of systemic retinoids within the past 3 months.
* Use of astringents, toners and skin cleansers for less than 2 weeks prior to the start of the study.
* Concomitant use of facial product containing glycolic or other acids, masks, washes or soaps containing benzoyl peroxide or salicylic acid, non mild cleansers or moisturizers containing retinol, salicylic or α- or β-hydroxy acids.
* Concomitant use of mega-doses of certain vitamins, such as vitamin D (>2000IU QD) vitamin B12, haloperidol, halogens such as iodide and bromide, lithium, hydantoin and phenobarbital.
* Facial procedures (chemical or laser peel, microdermabrasion, etc.) within the past 2 weeks or during the study.
* Concomitant use of tanning booths or sunbathing.
* Known hypersensitivity or previous allergic reaction to any of the active components, lincomycin, retinoids or excipients of the study product
* A significant medical history of or are currently immunocompromised
* Current drug or alcohol abuse. (Drug screening not required.)
* Use of any investigational therapy within 4 weeks of enrollment.
* Any other condition which, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1649 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- United States (27):
  - Radiant Research, Birmingham, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Center for Dermatology, Cosmetic and Laser Surgery, Fremont, California
  - University Clinical Trials, San Diego, California
  - Longmont Medical Research Network, Longmont, Colorado
  - FXM Research Corporation, Miami, Florida
  - FXM Research - Miramar, Miramar, Florida
  - Advanced Dermatolgy & Cosemtic Surgery, Ormond Beach, Florida
  - Dermatology Specialists, Louisville, Kentucky
  - Massachusettes General Hospital - Clinical Unit for Research Trials in Skin, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists, P.C., Omaha, Nebraska
  - Academic Dermatology Research, Albuquerque, New Mexico
  - Dermatology Research Associates, Inc., Cincinnati, Ohio
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Dermatology Associates of Knoxville, P.C., Knoxville, Tennessee
  - Tennessee Clinical Research, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - The Hair and Skin Research Treatment Center, Dallas, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Premier Clincial Research, Spokane, Washington
  - Advanced Healthcare, Milwaukee, Wisconsin
- Belize (2):
  - Dermatology And Skin Centre, Belize City
  - Dr. Moguel's Clinic, Belize City
- Canada (3):
  - K. Papp Clinical Research, Inc., Waterloo, Ontario
  - Windsor Clinical Research Center, Inc., Windsor, Ontario
  - Innovaderm Research, Inc., Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- CT Gel: Clindamycin 1% as clindamycin phosphate and tretinoin 0.025% (CT) applied topically to the face (including forehead, nose, cheeks, and chin) once daily in the evening for 12 weeks
- Clindamycin Gel: Clindamycin phosphate 1% applied topically to the face (including forehead, nose, cheeks, and chin) once daily in the evening for 12 weeks
- Tretinoin Gel: Tretinoin 0.025% applied topically to the face (including forehead, nose, cheeks, and chin) once daily in the evening for 12 weeks
- Vehicle Gel: Topical application to the face (including forehead, nose, cheeks, and chin) once daily in the evening for 12 weeks
Period: Overall Study
Arm/Group | CT Gel | Clindamycin Gel | Tretinoin Gel | Vehicle Gel
Started | 476 | 467 | 464 | 242
Completed | 414 | 416 | 405 | 211
Not Completed | 62 | 51 | 59 | 31
Not completed — Adverse Event | 6 | 0 | 5 | 0
Not completed — Lost to Follow-up | 26 | 19 | 17 | 11
Not completed — Lack of Efficacy | 1 | 2 | 2 | 2
Not completed — Non-Compliance with Study Treatment | 3 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 19 | 18 | 26 | 13
Not completed — Unable to Comply with Visit Schedule | 0 | 0 | 1 | 1
Not completed — Inclusion/Exclusion Criteria Not Met | 1 | 2 | 0 | 0
Not completed — Non-compliance with Treatment Regimen | 0 | 1 | 0 | 0
Not completed — Change/Discontinuation of Birth Control | 1 | 1 | 1 | 0
Not completed — Use of Prohibitive Medication | 2 | 1 | 3 | 0
Not completed — Pregnancy | 0 | 2 | 0 | 2
Not completed — Incarceration | 2 | 0 | 0 | 0
Not completed — Fear of Birth Defects | 0 | 0 | 1 | 0
Not completed — Transportation | 1 | 0 | 0 | 0
Not completed — Patient Withdrew from Study | 0 | 0 | 0 | 1
Not completed — Personal Reason | 0 | 1 | 0 | 0
Not completed — Dispensing Error | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT Gel | Clindamycin Gel | Tretinoin Gel | Vehicle Gel | Total
Number analyzed (Participants) | 476 | 467 | 464 | 242 | 1649
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (8.5) | 20.2 (8.1) | 20.2 (7.7) | 20.6 (8.4) | 20.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 266 | 264 | 153 | 952
  Male | 207 | 201 | 200 | 89 | 697
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 4 | 4 | 4 | 3 | 15
  Asian | 8 | 8 | 11 | 5 | 32
  Black | 94 | 85 | 103 | 51 | 333
  Multiracial | 12 | 16 | 19 | 5 | 52
  Native Hawaiian/Other Pacific Islander | 0 | 4 | 2 | 1 | 7
  White | 358 | 349 | 324 | 176 | 1207
  Missing | 0 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Lesion Counts (Total, Inflammatory, and Non-inflammatory) at Week 12 (End of Study)
Description: Acne lesion counts (inflammatory [papules, pustules, nodules], non-inflammatory [open and closed comedones], and total) were performed on the face of participants. Change from baseline is defined as Week 12 values minus Baseline values. The total lesion count is the sum of the inflammatory and non-inflammatory lesion counts.
Time Frame: Baseline, Week 12
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to and received at least one application of study product.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | CT Gel | Clindamycin Gel | Tretinoin Gel | Vehicle Gel
Number analyzed (Participants) | 476 | 467 | 464 | 242
lesions
  Inflammatory Lesion Counts | -15.5 (10.33) | -14.5 (9.37) | -13.9 (11.05) | -11.1 (11.70)
  Non-Inflammatory Lesion Counts | -23.2 (20.41) | -19.5 (19.72) | -22.1 (21.75) | -17.0 (20.58)
  Total Lesion Counts | -38.7 (26.80) | -34.0 (25.16) | -36.0 (28.26) | -28.1 (27.26)
Statistical Analysis 1: Comparison: CT Gel vs Clindamycin Gel; Test type: Superiority or Other; p = 0.063, Ranked ANCOVA — Inflammatory lesion count
Statistical Analysis 2: Comparison: CT Gel vs Tretinoin Gel; Test type: Superiority or Other; p = 0.003, Ranked ANCOVA — Inflammatory lesion count
Statistical Analysis 3: Comparison: CT Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA — Inflammatory lesion count
Statistical Analysis 4: Comparison: CT Gel vs Clindamycin Gel; Test type: Superiority or Other; p = 0.004, Ranked ANCOVA — Non-inflammatory lesion count
Statistical Analysis 5: Comparison: CT Gel vs Tretinoin Gel; Test type: Superiority or Other; p = 0.550, Ranked ANCOVA — Non-inflammatory lesion count
Statistical Analysis 6: Comparison: CT Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA — Non-inflammatory lesion count
Statistical Analysis 7: Comparison: CT Gel vs Clindamycin Gel; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA — Total lesion count
Statistical Analysis 8: Comparison: CT Gel vs Tretinoin Gel; Test type: Superiority or Other; p = 0.016, Ranked ANCOVA — Total lesion count
Statistical Analysis 9: Comparison: CT Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA — Total lesion count

2. Primary Outcome: The Percentage of Participants Who Had a Minimum 2-grade Improvement in the Investigator's Static Global Assessment (ISGA) Score From Baseline to Week 12
Description: The ISGA is a static ("snap-shot") evaluation of acne severity performed by an investigator/assessor at every visit. The ISGA score is measured on a 6-point ordinal scale, where 0=Clear and 5=Very Severe. Change is calculated as the Week 12 value minus the Baseline value.
Time Frame: Baseline, Week 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | CT Gel | Clindamycin Gel | Tretinoin Gel | Vehicle Gel
Number analyzed (Participants) | 476 | 467 | 464 | 242
percentage of participants | 36.3 | 26.6 | 26.1 | 20.2
Statistical Analysis 1: Comparison: CT Gel vs Clindamycin Gel; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — Data based on Data on File documenting FDA reanalysis request
Statistical Analysis 2: Comparison: CT Gel vs Tretinoin Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Data based on Data on File documenting FDA reanalysis request
Statistical Analysis 3: Comparison: CT Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Data based on Data on File documenting FDA reanalysis request

3. Secondary Outcome: Percent Change From Baseline in Lesion Counts (Inflammatory, Non-inflammatory, and Total) at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CT Gel | Clindamycin Gel | Tretinoin Gel | Vehicle Gel
Number analyzed (Participants) | 476 | 467 | 464 | 242
percent change
  Inflammatory Lesions | -60.5 (36.21) | -56.6 (44.99) | -54.5 (39.19) | -43.3 (44.9)
  Non-Inflammatory Lesions | -51.1 (33.02) | -42.9 (36.6) | -47.3 (43.5) | -36.0 (39.14)
  Total Lesions | -55.0 (30.47) | -49.0 (30.08) | -50.6 (34.82) | -39.1 (36.48)
Statistical Analysis 1: Comparison: CT Gel vs Clindamycin Gel; Test type: Superiority or Other; p = 0.065, Ranked ANCOVA — Inflammatory lesion count
Statistical Analysis 2: Comparison: CT Gel vs Tretinoin Gel; Test type: Superiority or Other; p = 0.002, Ranked ANCOVA — Inflammatory lesion count
Statistical Analysis 3: Comparison: CT Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA — Inflammatory lesion count
Statistical Analysis 4: Comparison: CT Gel vs Clindamycin Gel; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA — Non-inflammatory lesion count
Statistical Analysis 5: Comparison: CT Gel vs Tretinoin Gel; Test type: Superiority or Other; p = 0.284, Ranked ANCOVA — Non-inflammatory lesion count
Statistical Analysis 6: Comparison: CT Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA — Non-inflammatory lesion count
Statistical Analysis 7: Comparison: CT Gel vs Clindamycin Gel; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA — Total lesion count
Statistical Analysis 8: Comparison: CT Gel vs Tretinoin Gel; Test type: Superiority or Other; p = 0.028, Ranked ANCOVA — Total lesion count
Statistical Analysis 9: Comparison: CT Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA — Total lesion count

4. Secondary Outcome: The Percentage of Participants With a Subjects Global Assessment Score of 0 or 1 at Week 12
Description: The SGA score is a global evaluation of acne severity performed by participants at all visits and measured on a 5-point ordinal scale, where 0=My face is basically free of acne and 5=My face has blackheads and/or whiteheads. A score of 1=My face has several blackheads and/or whiteheads and small pimples, but there are no tender deep-seated bumps or cysts.
Time Frame: Week 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | CT Gel | Clindamycin Gel | Tretinoin Gel | Vehicle Gel
Number analyzed (Participants) | 476 | 467 | 464 | 242
participants | 62 | 60 | 62 | 50
Statistical Analysis 1: Comparison: CT Gel vs Clindamycin Gel; Test type: Superiority or Other; p = 0.671, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: CT Gel vs Tretinoin Gel; Test type: Superiority or Other; p = 0.919, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: CT Gel vs Vehicle Gel; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel

5. Secondary Outcome: The Percentage of Participants Who Had ISGA Scores of 0 or 1 at Week 12
Description: The ISGA is a static ("snap-shot") evaluation of acne severity performed by an investigator/assessor at every visit. The ISGA score is measured on a 6-point ordinal scale, where 0=Clear and 5=Very Severe. A score of 1=Skin Almost Clear: rare non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving and may be hyper-pigmented, though not pink-red) requiring no futher treatment in the Investigator's opinion.
Time Frame: Week 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | CT Gel | Clindamycin Gel | Tretinoin Gel | Vehicle Gel
Number analyzed (Participants) | 476 | 467 | 464 | 242
percentage of participants | 43.1 | 36.6 | 33.8 | 22.7
Statistical Analysis 1: Comparison: CT Gel vs Clindamycin Gel; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: CT Gel vs Tretinoin Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: CT Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Arm/Group | CT Gel | Clindamycin Gel | Tretinoin Gel | Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 1/476 | 1/467 | 3/464 | 1/242
Other Adverse Events (participants affected / at risk) | 27/476 | 34/467 | 27/464 | 18/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT Gel (N=476) | Clindamycin Gel (N=467) | Tretinoin Gel (N=464) | Vehicle Gel (N=242)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT Gel (N=476) | Clindamycin Gel (N=467) | Tretinoin Gel (N=464) | Vehicle Gel (N=242)
Nasopharyngitis (Infections and infestations) | 27 | 34 | 27 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.